CLINICAL TRIAL: NCT01034150
Title: Effects of Home-based Neurostimulation Associated With Motor Training in Chronic Stroke Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Adriana Bastos Conforto/ Staff neurologist, Hospital das Clinicas/University of Sao Paulo, Hospital das Clinicas/University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1309-06; 477916/06-6 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2009-12-11; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somatosensory stimulation (Active Comparator): Active group
  Interventions: Device: Relief band (Somatosensory stimulation)
- Control group (Placebo Comparator): Placebo stimulation
  Interventions: Device: Placebo stimulation

INTERVENTIONS:
Device: Relief band (Somatosensory stimulation) — Electrical median nerve stimulation
  Other Names: Relief band
  Arms: Somatosensory stimulation
Device: Placebo stimulation — Placebo stimulation
  Other Names: no stimulation
  Arms: Control group

SUMMARY:
Objective: To investigate effects of home-based somatosensory stimulation associated with motor training on improvement in performance of the paretic upper extremity in patients in the chronic phase after stroke.

DETAILED DESCRIPTION:
Design: Double-blind, randomized, controlled clinical trial. Setting: Home-based rehabilitation. Subjects: Patients in the chronic phase (> 6 months) after stroke. Interventions: Patients will be randomized to an active and a control group. In both groups, treatments will be performed at home, daily, over four weeks. Patients in the active group will be instructed to use a device that provides somatosensory stimulation in the form of electrical stimulation of the median nerve for two hours. Patients in the control group will also be instructed to use the device for two hours, and sham stimulation will be administered. In both groups, patients will be instructed to train activities with the paretic hand immediately after nerve stimulation.

Main measures: The primary outcome will be improvement in performance of the paretic hand evaluated by the Jebsen-Taylor test at end of treatment and four months after end of treatment, compared to baseline. Secondary outcomes were: 1) Compliance with the interventions, assessed through a daily written log, and oral reports of the patients; 2) safety profile of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years;
* single ischemic or hemorrhagic stroke in a cerebral hemisphere, documented by computed tomography (CT) or magnetic resonance imaging (MRI);
* stroke onset at least six months before;
* hand paresis with preserved ability to perform all tasks of the Jebsen-Taylor Test (JTT).

Exclusion Criteria:

* previous strokes;
* epilepsy and other neurological conditions;
* proprioceptive or tactile anesthesia;
* shoulder or hand pain;
* severe joint deformity;
* severe chronic disease;
* inability to give provide informed consent due to severe aphasia or cognitive impairment;
* left handedness before the stroke.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
the improvement in upper extremity performance assessed using Jebsen-Taylor test | Treatment lasted four weeks. Measures were performed before the treatment, immediately after the treatment and four months after the end of the treatment

SECONDARY OUTCOMES:
Compliance with the interventions, assessed through a daily written log, and oral reports of the patients | immediately after the treatment
Adverse events | at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Conforto, MD PhD, Principal Investigator — Hospital das Clínicas/FMUSP
Locations (1):
- University of São Paulo/General Hospital, São Paulo, São Paulo, Brazil